CLINICAL TRIAL: NCT01089751
Title: Efficacy of Sanctura XR (Trospium Chloride) for Reducing Overactive Bladder Symptoms in Female Subjects Refractory to Detrol LA (Tolterodine Tartrate Extended Release) Daily
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMA-SXR-09-004
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — trospium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sanctura XR® (Experimental): Sanctura XR® (trospium chloride) 60 mg once daily on an empty stomach for 14 weeks.
  Interventions: Drug: trospium chloride
- Placebo (Placebo Comparator): Placebo once daily on an empty stomach for 14 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: trospium chloride — Sanctura XR® (trospium chloride) 60 mg once daily on an empty stomach for 14 weeks
  Other Names: Sanctura XR®
  Arms: Sanctura XR®
Drug: placebo — Placebo once daily on an empty stomach for 14 weeks.
  Arms: Placebo

SUMMARY:
This study will investigate the safety and efficacy of Sanctura XR (trospium chloride) daily in reducing urgency, urinary frequency and urinary urge incontinence in female patients with incontinence refractory to Detrol LA (tolterodine tartrate extended release) 4 mg therapy.

ELIGIBILITY:
Inclusion Criteria:

* Taking Detrol® LA 4mg daily for a minimum of 1 month prior to Screening/Qualification
* Overactive Bladder syndrome with urgency, urinary frequency and urgency urinary incontinence
* Taking five or more concomitant medications (may be prescription, non-prescription, or supplement/vitamin) daily for indications other than Overactive Bladder (OAB).

Exclusion Criteria:

* Predominant stress or insensate incontinence
* History of neurogenic bladder
* Two urinary tract infections in the last six months
* Gastric by-pass (Roux-en-Y) surgery (adjustable gastric banding is allowed)
* Donated >500mL blood in the 30 days prior to the screening visit

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- La Mesa, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sanctura XR® | Placebo
Started | 163 | 159
Completed | 129 | 132
Not Completed | 34 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sanctura XR® | Placebo | Total
Number analyzed (Participants) | 163 | 159 | 322
Age Continuous [Mean (Full Range); unit: Years] | 56.3 [21 to 76] | 56.0 [21 to 84] | 56.1 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 159 | 322
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Continent (PPC)
Description: PPC is the percentage of patients with complete continence (without any urgency urinary incontinence episodes) during the 3-day bladder diary period associated with the Week 14 visit.
Time Frame: Week 14
Population: Modified intent-to-treat population included all randomized participants who were incontinent at Baseline with at least one urinary episode marked "Yes" for both Accidental leakage and Urgency associated void, and an Urgency severity rating ≥ 1 in the bladder diary.
Measure: Number; unit: Percentage of participants
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
Percentage of participants | 34.6 | 17.1

2. Secondary Outcome: Change From Baseline in Continent Days Per Week (CDW)
Description: Continent Days per Week is the average of the number of times an individual has no incontinence episodes in a day within the 3-day collection period calculated as 7 x (number of dry days within the 3-day diary period) divided by the number of valid diary days with at least one valid bladder diary entry during the 3-day period. A positive change from Baseline (more continent/fewer incontinent days per week ) indicated improvement.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Continent days per week
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
Continent days per week
  Baseline | 0.8 (1.46) | 1.0 (1.52)
  Change from Baseline at Week 14 | 2.6 (2.96) | 1.3 (2.73)

3. Secondary Outcome: Change From Baseline in Nocturic Toilet Voids
Description: A nocturic (nighttime) toilet void is identified if the patient marks "Yes" for both Toilet Voiding and Sleep Interruption in the 3-day bladder diary. The daily average number of nocturic toilet voids is obtained as the sum of all nighttime toilet voids over the 3-day bladder diary period divided by number of valid diary days with at least one valid bladder diary entry during the 3-day period. A negative change from Baseline (fewer nocturic toilet voids) indicated improvement.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nocturic toilet void
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
Nocturic toilet void
  Baseline | 2.2 (1.40) | 2.3 (1.41)
  Change from Baseline at Week 14 | -0.6 (1.51) | -0.3 (1.42)

4. Secondary Outcome: Change From Baseline in Urgency-Related Toilet Voids
Description: Urgency-related toilet void (or urinary urgency) is identified if the patient marks "Yes" for both Urgency Association Void and Toilet Voiding in the 3-day bladder diary. The daily average number of urgency-related voids is calculated as the sum of all urgency episodes over the 3-day bladder diary period divided by the number of valid diary days with at least one valid bladder diary entry during the 3-day period. A negative change from Baseline (fewer urgency related toilet voids) indicated improvement.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Toilet void
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
Toilet void
  Baseline | 7.6 (3.36) | 7.5 (3.62)
  Change from Baseline at Week 14 | -2.3 (3.78) | -1.6 (3.87)

5. Secondary Outcome: Change From Baseline in Daily Average Overactive Bladder-Symptom Composite Score (OAB-SCS)
Description: The OAB-SCS is derived from the 3-day bladder diary which includes: 1) 24-hour voiding frequency; 2) the Indevus Urgency Severity Scale (IUSS) Score (0=no urgency, 1=aware of urgency but is tolerable, 2=urgency discomfort interferes with activities/tasks, 3=extreme urgency discomfort that abruptly stops activities/tasks associated with each toilet void); and 3) the frequency of Urgency Urinary Incontinence episodes. Each toilet void is then assigned a point value from 1 (IUSS Score=0) to 5 (UUI episode not associated with a toilet void). The daily average OAB-SCS is then calculated based on the diary entries and assigned point values. The lowest possible daily average OAB-SCS is 0 (corresponding to no urgency in every void). There is no upper limit since the score is based on the number of voids per day. Scores <= 30 indicate mild OAB, scores > 30 to 39 indicate moderate OAB, and scores >= 40 indicate severe OAB. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
Score on a scale
  Baseline | 24.6 (9.07) | 23.7 (10.70)
  Change from Baseline at Week 14 | -6.5 (10.23) | -3.4 (11.44)

6. Secondary Outcome: Change From Baseline in Voided Volume
Description: Average volume of urine voided per toilet void is calculated by total volume collected in a 24-hour diary period divided by the number of individual entries of volume voided in that period. A positive change from Baseline (greater volume voided) indicated improvement. A negative change from Baseline (less volume voided) indicated a worsening.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeters (cc)
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
cubic centimeters (cc)
  Baseline | 183.5 (79.78) | 187.4 (78.76)
  Change from Baseline at Week 14 | 20.6 (89.62) | -8.0 (71.56)

7. Secondary Outcome: Change From Baseline in Urgency Severity
Description: The urgency severity per toilet void is based on the Indevus Urgency Severity Scale (IUSS). The patient recorded urinary urgency severity in a 3-day bladder diary using a 4-point scale: 0=None-no urgency (best), 1=Slight-aware of urgency but is tolerable, 2=Moderate-urgency discomfort interferes with activities/tasks, 3=Severe-extreme urgency discomfort that abruptly stops activities/tasks (worst). Urgency Severity is calculated as the sum of all IUSS scores during the 3-day diary period divided by the number of toilet voids recorded during that period. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
Score on a scale
  Baseline | 1.4 (0.60) | 1.3 (0.56)
  Change from Baseline at Week 14 | -0.4 (0.67) | -0.3 (0.60)

8. Secondary Outcome: Change From Baseline in Urgency Urinary Incontinence (UUI)
Description: Urgency urinary incontinence is identified if the patient marks "Yes" for both Accidental Leakage and Urgency Associated Void in the 3-day bladder diary, and the Urgency Severity score is ≥ 1. Average daily episodes of UUI is calculated as the sum of all UUI episodes over 3-day diary period divided by the number of valid diary days with at least one valid bladder diary entry during the 3-day period. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: UUI episodes
Arm/Group | Sanctura XR® | Placebo
Number analyzed (Participants) | 156 | 152
UUI episodes
  Baseline | 2.9 (2.99) | 3.0 (2.72)
  Change from Baseline at Week 14 | -1.1 (2.24) | -0.6 (2.22)

ADVERSE EVENTS:
Description: The safety population (all participants who took at least 1 dose of study medication) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Sanctura XR® | Placebo
Serious Adverse Events (participants affected / at risk) | 2/162 | 3/158
Other Adverse Events (participants affected / at risk) | 20/162 | 8/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sanctura XR® (N=162) | Placebo (N=158)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sanctura XR® (N=162) | Placebo (N=158)
Dry mouth (Gastrointestinal disorders) | 11 | 6
Constipation (Gastrointestinal disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.